CLINICAL TRIAL: NCT06789211
Title: Impact of Symptoms and Left Ventricular Systolic Function in Patients With Moderate Mixed Aortic Valve Disease
Brief Title: Outcomes in Moderate Mixed Aortic Valve Disease
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Edwards Lifesciences (Industry); Queen Mary Hospital, Hong Kong (Other); National Heart Centre Singapore (Other); Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Nina Ajmone Marsan, MD, PhD, Leiden University Medical Center
Other Study IDs: DAP/tak/1662024; THV-I24-181 (Other: Edwards Lifesciences)
Record Dates: First submitted 2025-01-15; First posted 2025-01-23 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-01

CONDITIONS: Mixed Aortic Valve Disease
Keywords: valvular heart disease; mixed aortic valve disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Moderate Mixed Aortic Valve Disease
- Severe Aortic Stenosis
- Severe Aortic Regurgitation

SUMMARY:
Mixed aortic valve disease (MAVD) is defined as the combination of aortic valve stenosis (AS) and regurgitation (AR) and is relatively frequent, with a reported prevalence up to 20-30% of patients with aortic valve disease. Mortality of patients with moderate MAVD (coexistence of both moderate AS and moderate AR) is largely unknown, and therefore there are currently no guidelines-based indications for surgical or transcatheter intervention for these patients, which is considered only when one of the two lesions (AS or AR) becomes severe. Of note, indication for valve intervention in patients with isolated moderate AS is currently under investigation in several randomized clinical trials but only in the presence of relevant symptoms and signs of left ventricular (LV) dysfunction. One initial single-center study including 250 patients with moderate MAVD has evaluated outcomes in this specific subgroup and showed that patients with asymptomatic moderate MAVD and preserved left ventricular ejection fraction (LVEF) had similar adverse event rates (progression to New York Heart Association (NYHA) class III-IV, aortic valve intervention or cardiac death) to patients with isolated asymptomatic severe AS with preserved LVEF. However, the results were primarily driven by the progression of the NYHA Class and aortic valve replacement, and larger multi-center studies are advocated to confirm these findings, which may therefore identify a (new) group of high risk patients who should in principle benefit from an aortic valve intervention as much as patients with isolated severe AS. In addition, prognostic factors (including clinical and echocardiographic characteristics) for risk-stratification of patients with moderate MAVD have not been identified, which may help to refine the indication for valve intervention and optimize patient management.

DETAILED DESCRIPTION:
Hypothesis: Patients with moderate MAVD may have similar mortality rates compared to patients with isolated severe AS or severe AR and therefore benefit from aortic valve intervention. The presence of symptoms or impaired LV function may further identify a higher risk group together with other clinical or echocardiographic parameters.

Objectives:

1. To compare mortality rates in patients with moderate MAVD to isolated severe AS and isolated severe AR in a multi-center setting, adjusting for potential differences in clinical and echocardiographic variables and for the occurrence of aortic valve intervention.
2. To identify clinical and echocardiographic characteristics associated with increased mortality in this specific population and potentially propose dedicated risk scoring and adjusted cut-off values for the various parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with concomitant moderate AS and moderate AR
2. Patients with isolated severe AS
3. Patients with isolated severe AR

Exclusion Criteria:

1. Previous aortic valve surgery
2. Concomitant left valvular heart disease more than mild grade
3. Acute AR
4. Bad echocardiographic image quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with concomitant moderate AS and moderate AR, patients with isolated severe AS and isolated severe AR.
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 2003-2024

SECONDARY OUTCOMES:
All-cause mortality or aortic valve replacement | 2003-2024

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No